CLINICAL TRIAL: NCT00236002
Title: A Phase III, Double-blind, Randomized, Parallel Group, Placebo-controlled Study of Oral Fosamax, 70 mg Once a Week, for the Prevention of Androgen Deprivation Bone Loss in Non-metastatic Prostate Cancer
Brief Title: Cancer and Osteoporosis Research With Alendronate and Lupron (C.O.R.A.L )
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow accrual than anticipated.
Sponsor: Canadian Urology Research Consortium (Other)
Collaborators: Abbott (Industry); Merck Frosst Canada Ltd. (Industry)
Responsible Party: Dr. Laurence Klotz, Canadian Urology Research Consortium
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ACA-CANA-04-012
Record Dates: First submitted 2005-10-11; First posted 2005-10-12 (Estimated); Last update posted 2009-08-12 (Estimated); Status verified 2009-08

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Alendronate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- placebo (Placebo Comparator)
  Interventions: Drug: Alendronate

INTERVENTIONS:
Drug: Alendronate — Alendronate 70mgm once a week for one year
  Other Names: fosamax

SUMMARY:
Multi-center,double blind randomized phase III placebo controlled study in 250 men with histologically proven prostate cancer with out bone metastases who are beginning ADT therapy and who will receive concomitant treatment with either oral Fosamax 70mg once weekly or placebo for one year.These men will be treated and follow up for one year,during which time changes in BMD, markers of bone resorption and formation will be monitored.All patients will receive calcium and vitamin D through out the study.

DETAILED DESCRIPTION:
This is a phase three multicentre, double blind, randomize parallel group, placebo-controlled study in 250 men with histologically proven cancer without bone metastases who are beginning ADT therapy and who will receive a concomitant treatment with either oral Fosamax 70 mg once a weak (n=125) or placebo (n=125) for one year. Changes in BMD, markers of bone absorption and formation are monitored.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically proven, non-metastatic (M0) adenocarcinoma of the prostate.
* Life expectancy of > 12 months.
* Initiation of treatment with the luteinizing hormone-releasing hormone agonist (LHRH-a) Lupron no more than 15 days prior or 30 days following, baseline visit.
* Requiring treatment with LHRH agonists for prostate cancer, for a duration of at least 12 months from baseline.
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2
* Prior to any study-specific procedures, subject (and/or their legally authorized representative) has voluntarily signed and dated an informed consent form.

Exclusion Criteria:

Bone Metastases Current or previous use with in past 12 months of bisphosphonate. Known hypersensitivity to LHRH. Hypocalcaemia. Severe renal impairment, Abnormal liver function, Hypothyroidism, Hyperthyroidism, Bilateral hip replacement.

Use of LHRH or anti-androgen medication within last 12 months. Abnormalities of esophagus which delay esophageal emptying. Inability to stand or sit upright for at least 30 minutes.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2005-07; Primary Completion 2007-11 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Bone mineral density | ONE YEAR

SECONDARY OUTCOMES:
Blood and urine to check liver,kidney,thyroid functions. PSA and bone markers will also be checked | every 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Lesley Carr, M.D., Principal Investigator — Sunnybrook Health Sciences Centre